CLINICAL TRIAL: NCT02270840
Title: Effect of Biventricular Upgrade on Left Ventricular Reverse Remodeling and Clinical Outcomes in Patient With Left Ventricular Dysfunction and Intermittent or Permanent Apical/Septal Right Ventricular Pacing (Budapest CRT Upgrade Study)
Brief Title: Budapest Upgrade CRT Study (Version 009-4.1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University Heart and Vascular Center (Other)
Collaborators: University of Rochester (Other); Sheba Medical Center (Other Government); Pharmahungary Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Budapest Upgrade CRT 009-4.1
Record Dates: First submitted 2014-10-17; First posted 2014-10-21 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Cardiomyopathy
Keywords: cardiac resynchronization therapy
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT-D (Active Comparator): Patients currently implanted with a single or dual chamber pacemaker or ICD will be upgraded to CRT.
  Interventions: Device: CRT-D
- Only ICD (No Intervention): In the ICD arm, choosing single or dual chamber device is based upon the investigator's discretion.
  Subjects meeting the inclusion criteria (and if exclusion criteria are not present) patients will be randomized to CRT-D upgrade or ICD only (either continued ICD therapy in patients currently implanted with a defibrillator or implantation of a defibrillator in eligible patients who are currently implanted with pacemaker-only).

INTERVENTIONS:
Device: CRT-D — Biventricular upgrade. Subjects meeting the inclusion criteria (and if exclusion criteria are not present) patients will be randomized to CRT-D upgrade or ICD only (either continued ICD therapy in patients currently implanted with a defibrillator or implantation of a defibrillator in eligible patients who are currently implanted with pacemaker-only).
  Arms: CRT-D

SUMMARY:
Effect of biventricular upgrade on left ventricular reverse remodeling and clinical outcomes in patient in left ventricular dysfunction and intermittent or permanent apical/septal right ventricular pacing (Budapest CRT upgrade study)

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of upgrade to a CRT-D device on clinical and echocardiographic response at 12-month in patients with left ventricular dysfunction (LVEF ≤35%), symptomatic heart failure (NYHA II, III, IV-a), and intermittent or permanent right ventricular pacing with paced QRS complex ≥ 150 ms compared to continued therapy with a single or dual chamber pacemaker (PM) or ICD.

Prospective, post-market, international multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over the age of 18 (expected survival time: over 1 year)
* Patients with ischemic or non-ischemic cardiomyopathy;
* Those implanted with a single or dual chamber ICD or implanted with a single or dual chamber pacemaker at least 6 months before inclusion;
* Elective generator replacement or upgrade from pacemaker-only to ICD therapy may be indicated at the time of enrollment, but are not required;
* Right ventricular pacing 20-100% in at least the last 90 days before enrollment (with an optimal AV interval based on the physician's discretion to avoid unnecessary right ventricular stimulation);
* Symptomatic heart failure for at least 3 months before inclusion;
* NYHA functional class II or III, or IV a;
* Left ventricular ejection fraction measured by echocardiography ≤ 35%;
* Paced QRS complex ≥ 150 ms;
* Optimal heart failure medical therapy;
* Informed consent obtained.

Exclusion Criteria:

* Intrinsic QRS with LBBB morphology (measured at VVI 40 bpm setting as per protocol);
* CABG or PCI in the past 3 months;
* Acute myocardial infarction in the past 3 months;
* Unstable angina;
* Planned coronary revascularization (PCI or CABG);
* Planned cardiac transplantation;
* Acute myocarditis;
* Infiltrative myocardial disease;
* Hypertrophic cardiomyopathy;
* Severe primary mitral and aortic valve stenosis or regurgitation;
* Women who are pregnant or plan to become pregnant or breastfeeding;
* Subjects who are unable or unwilling to cooperate with the study protocol;
* Tricuspid valve prosthesis;
* Any serious disease likely to interfere with the conduct of the study;
* Participation in other clinical trial;
* Patients geographically not stable or unavailable for follow-up;
* Chronic, severe renal dysfunction (creatinine value > 200 μmol/l);
* Severe RV dilatation (RV basal diameter >50mm);
* Severe tricuspid insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
A composite clinical and echocardiographic end point comprising the first occurrence of a non-fatal heart failure event, all-cause mortality, or < 15% reduction in echocardiography determined LVESV from baseline to 12-month. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, Study Director — University of Rochester Medical Center, Rochester, NY, USA; Ilan Goldenberg, Prof. MD, Study Director — Sheba Medical Center; Béla Merkely, Prof. MD, Principal Investigator — Semmelweis University Hearth and Vascular Center, Budapest, Hungary; Annamaria Kosztin, MD, Study Director — Semmelweis University Hearth and Vascular Center, Budapest, Hungary
Locations (17):
- Germany (2):
  - Hannover Medical School, Hanover
  - Herzzentrum Leipzig GmbH, Leipzig
- Hungary (6):
  - Second Department of Internal Medicine and Cardiology Center, Faculty of Medicine, University of Szeged, Szeged, Csongrád megye
  - Institute of Cardiology University of Debrecen, Debrecen, Hajdú-Bihar
  - Hungarian Institute of Cardiology, Budapest
  - Semmelweis University Heart and Vascular Center, Budapest
  - Depratment of Cardiology, Military Hospital, Hungarian Army Medical Center, Budapest
  - University of Pécs Medical School, Heart Institute, Pécs
- Israel (2):
  - Barzilai Medical Center, Ashkelon
  - Kaplan Medical Center, Rehovot
- Poland (4):
  - Central Clinical Hospital of Silesia, Department of Electrocardiology, Katowice
  - Department of Interventional Cardiology, Medical University of Lodz,, Lodz
  - Medical Center Tronik, Lodz
  - Medical University of Warsaw, Warsaw
- Clinical Center of Serbia, Belgrade, Serbia
- SK-01 National Institute for Cardiovascular Diseases, Bratislava, Slovakia
- University Medical Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Merkel E, Hatala R, Szigeti M, Schwertner W, Lakatos B, Behon A, Goscinska-Bis K, Milasinovic G, Papp R, Ruppert M, Saghy L, Clemens M, Solomon SD, Kutyifa V, Kovacs A, Kosztin A, Merkely B. Upgrading Right Ventricular Pacing to Cardiac Resynchronization in HFrEF Patients Improves Symptoms and Functional Outcomes. JACC Heart Fail. 2025 Feb;13(2):265-273. doi: 10.1016/j.jchf.2024.09.011. Epub 2024 Nov 27. PMID 39614838
- [Derived] Merkely B, Geller L, Zima E, Osztheimer I, Molnar L, Foldesi C, Duray G, Wranicz JK, Nemeth M, Goscinska-Bis K, Hatala R, Saghy L, Veres B, Schwertner WR, Fabian A, Fodor E, Goldenberg I, Kutyifa V, Kovacs A, Kosztin A. Baseline clinical characteristics of heart failure patients with reduced ejection fraction enrolled in the BUDAPEST-CRT Upgrade trial. Eur J Heart Fail. 2022 Sep;24(9):1652-1661. doi: 10.1002/ejhf.2609. Epub 2022 Jul 22. PMID 35791276
- [Derived] Merkely B, Kosztin A, Roka A, Geller L, Zima E, Kovacs A, Boros AM, Klein H, Wranicz JK, Hindricks G, Clemens M, Duray GZ, Moss AJ, Goldenberg I, Kutyifa V. Rationale and design of the BUDAPEST-CRT Upgrade Study: a prospective, randomized, multicentre clinical trial. Europace. 2017 Sep 1;19(9):1549-1555. doi: 10.1093/europace/euw193. PMID 28339581
- See also: Rationale and design of the BUDAPEST-CRT Upgrade Study: a prospective, randomized, multicentre clinical trial — https://pubmed.ncbi.nlm.nih.gov/28339581/